CLINICAL TRIAL: NCT02550210
Title: A Study to Evaluate the Accuracy of a Breast Cancer Locator (BCL) in Patients With Palpable Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., MD, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D15120
Record Dates: First submitted 2015-08-25; First posted 2015-09-15 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast Conserving Surgery; Breast Imaging; Breast Diagnostics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Breast Cancer Locator (BCL) (Experimental): The Breast Cancer Locator (BCL) uses 3D printing to create a bra-like plastic form that matches the breast surface when the patient is in the supine MRI (and surgical) position. This locator will be constructed pre-operatively, sterilized and provided to the surgeon at the time of procedure.
  Interventions: Device: Breast Cancer Locator (BCL)

INTERVENTIONS:
Device: Breast Cancer Locator (BCL) — This locator is constructed pre-operatively, sterilized and provided to the surgeon at the time of the procedure. The outline of the breast cancer on the breast surface at the point where the cancer is closest to the skin is built into the locator, so that the surgeon can simply apply the locator to the patient's breast and trace the tumor outline on the skin.

SUMMARY:
In this study, the investigators will enroll women with palpable cancers to assess the accuracy of the Breast Cancer Locator (BCL) and the concomitant procedure as a vehicle to optimize and validate the approach in such surgical cases. This approach of adopting palpable cancer patients before initiating an evaluative trial of the BCL in non-palpable breast cancer cases ensures that the BCL does not substantially alter or modify the standard-of-care procedure.

DETAILED DESCRIPTION:
The investigators propose to test whether the Breast Cancer Locator (BCL) accurately defines the edges of the tumor. Twenty patients with palpable invasive breast cancer will undergo preoperative supine MRI, the creation of a BCL, and breast-conserving surgery using the BCL as an adjunct to palpation-guided tumor resection. Participants will also have the tumor position on their skin localized with the supine MR/optical scan/tracker method. The primary objective is to measure the distance from the center of the spots made by the BCL to the cancer edges.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histologic diagnosis of palpable invasive breast cancer or ductal carcinoma in situ
* Patient desire to undergo breast surgery
* Ability to voluntarily provide informed consent to participate prior to any study-related assessments/procedures being conducted
* The cancer enhances on breast MRI imaging.

Exclusion Criteria:

* Absolute contraindication to MRI, including presence of implanted electrical device (pacemaker or neurostimulator), aneurysm clip, or metallic foreign body in or near eyes
* Severe claustrophobia
* Contraindication to use of gadolinium-based intravenous contrast, including life-threatening allergy or compromised renal function (creatinine > 2.0)
* History of median sternotomy
* Pregnancy. Patient attestation that they are not pregnant will be acceptable as per standard policy for MRIs at DHMC.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Cancer Locator (BCL): The Breast Cancer Locator (BCL) uses 3D printing to create a bra-like plastic form that matches the breast surface when the patient is in the supine MRI (and surgical) position. This locator will be constructed pre-operatively, sterilized and provided to the surgeon at the time of the procedure.
  Breast Cancer Locator (BCL): This locator is constructed pre-operatively, sterilized and provided to the surgeon at the time of the procedure. The outline of the breast cancer on the breast surface at the point where the cancer is closest to the skin is built into the locator so that the surgeon can simply apply the locator to the patient's breast and trace the tumor outline on the skin.
Period: Overall Study
Arm/Group | Breast Cancer Locator (BCL)
Started | 23
Completed | 19
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Breast Cancer Locator (BCL)
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years] | 59 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: The Distance Measured by Pathology From the Tumor Edge to the Center of the Ink Spots, as Marked by the Black Inked Pins.
Description: Five measurements will be made per patient and the mean difference in distance will be derived between the palpated and the co-registered supine MRI-optical scan image predicted tumor edges. The BCL will be considered accurate if all 5 measurements are > 0 cm from the tumor edge.
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Breast Cancer Locator (BCL)
Number analyzed (Participants) | 18
cm | 1.7 (1.2)

2. Secondary Outcome: Positive Margin Rate
Description: The positive margin rate as defined by standard pathologic evaluation of the entire specimen.
Time Frame: 30 Days
Measure: Number; unit: percentage
Arm/Group | Breast Cancer Locator (BCL)
Number analyzed (Participants) | 19
percentage | 0

3. Secondary Outcome: The Distances Between the Specimen Edges as Determined by the Breast Cancer Locator and by the Supine MRI/Optical Scan/ Tracker System
Description: Distances will be measured and descriptive statistics will be employed.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Breast Cancer Locator (BCL)
Number analyzed (Participants) | 19
cm | 0.33 (0.32)

4. Secondary Outcome: Mean Resection Specimen Volume
Description: Volumes will be measured and descriptive statistics will be employed. The specimen volume is determined by recording the water displacement and specimen scanning.
Time Frame: 30 days from surgery
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Breast Cancer Locator (BCL)
Number analyzed (Participants) | 19
cm3 | 116 (73)

ADVERSE EVENTS:
Time Frame: From the inception of baseline to end of intervention: 5 years
Description: Regular investigator assessment and regular laboratory testing
Arm/Group | Breast Cancer Locator (BCL)
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02550210/Prot_SAP_000.pdf